CLINICAL TRIAL: NCT07106398
Title: The Effectiveness of rTMS on Improving Food Craving and Weight Control in Adults Without Serious Mental Illness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Cheng Pak Wing, Calvin, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 25-282
Record Dates: First submitted 2025-07-21; First posted 2025-08-06 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Food Cravings; rTMS
Keywords: rtms; food cravings; healthy adults
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy adults (Experimental): Healthy adults aged 18-65 Self-reported food craving or weight control issues
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — Six sessions of rTMS using the EXOMIND™ device, administered once or twice a week.
  Each session will deliver 6,300 pulses at alternating frequencies of 12, 15, and 18 Hz, with a total duration of 24 minutes and 30 seconds.
  The target site would be left dorsolateral prefrontal cortex (DLPFC), determined by the most common used 5-cm rule. The procedure would be conducted in the research centre with medical staff supported.

SUMMARY:
Department of Psychiatry | Li Ka Shing Faculty of Medicine

The University of Hong Kong

The Effectiveness of rTMS on Improving Food Cravings and Weight Control

in Adults without Serious Mental Illness

Introduction

The investigators would like to invite participants to participate in an observational study on the efficacy of using magnetic fields to improve food cravings and weight control in adults without serious mental illness.

The research leader is Dr. Cheng Pak Wing, Assistant Professor, Department of Psychiatry, Queen Mary Hospital/HKU Li Ka Shing Faculty of Medicine.

Please read the following information carefully. If necessary, participants can discuss it with relatives, friends or doctors. If anything is unclear, or if participants would like more information, please ask us. Please carefully consider whether participants are willing to participate in this research.

Research Purpose

Food cravings are a common experience that can significantly impact an individual's mental and physical health. These intense desires for specific foods often lead to overconsumption of unhealthy foods, contributing to obesity, poor nutritional intake, and associated health conditions. Understanding the neural mechanisms behind food cravings is crucial for developing effective interventions to manage them.

rTMS is a non-invasive brain stimulation technique that uses magnetic fields to modulate neural activity in targeted brain regions. Over the years, rTMS has shown promise in treating various mental health conditions, including depression, obsessive-compulsive disorder (OCD) and eating disorders.

Research Methods

Participants

Healthy adults aged 18-65 with self-reported food cravings or weight control issues.

Treatment protocol

Six sessions of rTMS using the EXOMIND™ device, administered once or twice a week.

Each session will deliver 6,300 pulses at alternating frequencies of 12, 15, and 18 Hz, with a total duration of 24 minutes and 30 seconds.

The target site would be left dorsolateral prefrontal cortex (DLPFC), determined by the most common used 5-cm rule. The procedure would be conducted in the research centre with medical staff supported.

A checklist of potential adverse effects from TMS administration will be referenced from existing literature to monitor tolerability and adverse events during each session. Blood pressure and heart rate will be recorded at the beginning and end of each session.

Assessment

Participants will be assessed at three time points: baseline (pre-intervention), post-intervention, and four weeks post-intervention.

Assessments: Food Cravings Questionnaire-Trait (FCQ-T), Perceived Stress Scale (PSS), Patient Health Questionnaire-9 (PHQ-9), and BMI.

Demographics: Age, gender, years of education, place of birth, marital status, number of children, financial condition, household income, family history of eating problems will be collected upon study entry. Medical history in relation to mental illnesses and medications will also be assessed.

DETAILED DESCRIPTION:
Risks of Participation

Participants may experience mild discomfort from brain stimulation treatment. A small percentage of users may experience dizziness, headache, or nausea. The side effects of brain pulse stimulation therapy are short-lived and are not known to cause any permanent damage. If participants feel unwell after completing the brain pulse stimulation treatment, please inform the staff and therapist.

Note: Patients who have had metal implants in the head, neck, or upper back, or who have had metal teeth/dental trays or pacemakers, should not receive brain stimulation.

Benefits of Participation

The investigators sincerely invite participants to participate in this study. The valuable information participants provide will help us understand the effect of using magnetic fields to improve food cravings or weight control issues in adults. All procedures involved in the study are provided free of charge.

Voluntary Participation

Participation in our research is entirely voluntary, and participants have the right to withdraw from research at any time. Participants' decision to participate in or withdraw from the study will not affect participants' existing treatment or services. The information participants provide will be kept strictly confidential and all information will be used for research purposes only.

Financial Costs

Participants will not be charged for the service. Study article will not be continued to be available to subjects after the study until it is commercially available.

Confidentiality of Information

Any information about participants obtained during the research process will be kept strictly confidential. Personal data will be kept for 5 years after completion of study and publications, and will be destroyed after completion of publications. Any information about participants that is released outside the hospital (e.g. in scientific literature or reports) will not have personally identifiable information about participants. Each study participant has the right to access their personal data and publicly reported study results if required, and participants' contact details will be reserved for future follow-up studies.

Under the laws of Hong Kong (especially the Personal Data (Privacy) Ordinance, Cap. 486), participants have the right to keep participants' personal data confidential, such as the collection of personal data in or in connection with this research, safeguard, retain, manage, control, use (analyse or compare), transfer within or outside Hong Kong, non-disclosure, erasure and/or deal within any way. If participants have any questions, participants can consult the Office of the Privacy Commissioner for Personal Data or call its office (telephone number: 2827 2827) to properly supervise or monitor the protection of participants' personal data so that participants are fully aware and aware of ensuring compliance with the law to protect private data meaning.

By agreeing to participate in this study, participants expressly authorize:

To oversee this study, authorize the principal investigator and his research team and the Institutional Review Board of the University of Hong Kong / Hospital Authority Hong Kong West Cluster to obtain, use and retain participants in the manner specified in this study and this informed consent, and

Authorize relevant government agencies (such as the Hong Kong Department of Health) to obtain participants' personal data to check and verify the integrity of the research data and assess the consistency of the research agreement with the relevant requirements.

Enquiries

This study has been reviewed and approved by the Institutional Review Board of the University of Hong Kong/ Hospital Authority Hong Kong West Cluster. If participants are willing to participate in the research, please sign the enclosed informed consent form and keep this fact sheet for reference.

The study was coordinated by Dr. Cheng Pak Wing, Assistant Professor, Department of Psychiatry, Faculty of Medicine, The University of Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Aged between 18-65
* Self-reported food craving or weight control issues

Exclusion Criteria:

* People with serious mental illness
* Severe neurological conditions
* Contraindications for rTMS
* People on weight-reduction medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2027-06-27 (Estimated); Study Completion 2028-06-27 (Estimated)

PRIMARY OUTCOMES:
Food Cravings Questionnaire-Trait (FCQ-T) | Baseline: 1-week before rTMS intervention starts Post-intervention: 1-week after the last session of rTMS intervention 4-week post-intervention: 4-week after the last session of rTMS intervention
  Using Food Cravings Questionnaire-Trait (FCQ-T) to measure level of food cravings.
  The questionnaire consists of 23 questions, participants are required to rate the frequency of each statement with a 6-likert scale. By summing up the scores of the scles, higher scores represent higher level of food cravings.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | Baseline: 1-week before rTMS intervention starts Post-intervention: 1-week immediately after the last session of rTMS intervention 4-week post-intervention: 4-week after the last session of rTMS intervention
  Using perceived stress scale (PSS) to evaluate perceived stress levels.
  First, reverse the scores for questions 4, 5, 7, and 8. On these 4 questions, change the scores like this: 0 = 4, 1 = 3, 2 = 2, 3 = 1, 4 = 0.
  Now add up the scores for each item to get a total. The total score is ___________.
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress
Patient Health Questionnaire-9 (PHQ-9) | Baseline: 1-week before rTMS intervention starts Post-intervention: 1-week immediately after the last session of rTMS intervention 4-week post-intervention: 4-week after the last session of rTMS intervention
  Using Patient Health Questionnaire-9 (PHQ-9) to assess depressive symptoms
  Scoring: add up all checked boxes on PHQ-9 (For every 3 Not at all = 0; Several days = 1; More than half the days = 2; Nearly every day = 3)
  Interpretation of Total Score: Total Score Depression Severity 1-4: Minimal depression 5-9: Mild depression 10-14: Moderate depression 15-19: Moderately severe depression 20-27: Severe depression
BMI | Baseline: the day the rTMS intervention starts Post-intervention: the day the last session rTMS intervention
  Using BMI to measure the objective weight changes in between pre and post intervention.
  To calculate Body Mass Index (BMI), divide participants' weight in kilograms by the square of participants' height in meters

CONTACTS AND LOCATIONS:
Locations (1):
- Sassoon Road Campus, HKU, Hong Kong, Pok Fu Lam, Hong Kong

IPD SHARING:
Plan to Share IPD: No
protecting participant data

REFERENCES:
- [Background] Dalton B, Maloney E, Rennalls SJ, Bartholdy S, Kekic M, McClelland J, Campbell IC, Schmidt U, O'Daly OG. A pilot study exploring the effect of repetitive transcranial magnetic stimulation (rTMS) treatment on cerebral blood flow and its relation to clinical outcomes in severe enduring anorexia nervosa. J Eat Disord. 2021 Jul 9;9(1):84. doi: 10.1186/s40337-021-00420-w. PMID 34243816
- [Background] Fitzsimmons SMDD, van der Werf YD, van Campen AD, Arns M, Sack AT, Hoogendoorn AW; other members of the TETRO Consortium; van den Heuvel OA. Repetitive transcranial magnetic stimulation for obsessive-compulsive disorder: A systematic review and pairwise/network meta-analysis. J Affect Disord. 2022 Apr 1;302:302-312. doi: 10.1016/j.jad.2022.01.048. Epub 2022 Jan 15. PMID 35041869
- [Background] Voineskos D, Blumberger DM, Rogasch NC, Zomorrodi R, Farzan F, Foussias G, Rajji TK, Daskalakis ZJ. Neurophysiological effects of repetitive transcranial magnetic stimulation (rTMS) in treatment resistant depression. Clin Neurophysiol. 2021 Sep;132(9):2306-2316. doi: 10.1016/j.clinph.2021.05.008. Epub 2021 Jun 1. PMID 34167891
- [Background] Sabe M, Hyde J, Cramer C, Eberhard A, Crippa A, Brunoni AR, Aleman A, Kaiser S, Baldwin DS, Garner M, Sentissi O, Fiedorowicz JG, Brandt V, Cortese S, Solmi M. Transcranial Magnetic Stimulation and Transcranial Direct Current Stimulation Across Mental Disorders: A Systematic Review and Dose-Response Meta-Analysis. JAMA Netw Open. 2024 May 1;7(5):e2412616. doi: 10.1001/jamanetworkopen.2024.12616. PMID 38776083

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT07106398/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT07106398/ICF_001.pdf